CLINICAL TRIAL: NCT00262314
Title: Prospective, Open-label Tolerability and Safety Monitoring Study of Novantrone in a Selected Cohort of Multiple Sclerosis Patients
Acronym: RENEW
Status: Completed | Type: Observational
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Other Study IDs: 24293; 19-297; NCT00016614 (obsolete NCT alias)
Record Dates: First submitted 2005-12-05; First posted 2005-12-06 (Estimated); Results first posted 2010-06-23 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-10

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The overall objective of this study is to collect data relevant to the tolerability of Novantrone® therapy in patients with multiple sclerosis (MS) using dosing and monitoring recommendations specified in the package insert.

DETAILED DESCRIPTION:
This phase IV, multicenter, prospective, open-label tolerability and safety monitoring study will enroll a select cohort of 500 multiple sclerosis patients receiving commercially available Novantrone®. The patients will be assessed every 3 months during treatment followed by annual assessment for a total of five (5) years.

The select cohort of MS patients enrolled will have secondary (chronic) progressive, progressive relapsing, or worsening relapsing-remitting disease (i.e., patients whose neurological status is significantly abnormal between relapses).

The overall objective of this study is to collect data relevant to the tolerability of Novantrone® therapy in patients with multiple sclerosis (MS) using dosing and monitoring recommendations specified in the package insert.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for inclusion into this study, the subjects must fulfill all of the following criteria:
* Platelet count >100,000 cells/µL
* Granulocyte count > 2000 cells/µL
* Age 18-65 years
* Negative pregnancy test for female patients who are biologically capable of becoming pregnant, even if they are taking birth control
* For patients of reproductive age, agreement to practice effective contraception throughout the study and for 6 months following the last administration of Novantrone®
* Signed Inform Consent.

Exclusion Criteria:

* To be eligible for inclusion in this study the subjects must not meet any of the following criteria:
* Presence of cardiac risk factors:
* History of congestive heart failure
* LVEF < 50% determined by echocardiography or MUGA
* Previous treatment with Novantrone®, other anthracenediones, or anthracyclines
* Prior mediastinal radiotherapy or total lymphoidal irradiation
* AST, ALT, bilirubin > 2x upper limits of normal
* Severe untreated infection (including current urinary tract infection)
* Nursing or pregnant women)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients with a clinically definite or laboratory supported diagnosis of MS and having secondary (chronic) progressive, progressive relapsing, or worsening relapsing-remitting disease (i.e., patients whose neurologic status is significantly abnormal between relapses). Patients with primary progressive disease will not be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 509 (Actual)
Dates: Start 2000-10; Primary Completion 2008-01 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randy Bennett, Study Director — EMD Serono
Locations (1):
- Registrat Inc, Lexington, Kentucky, United States

REFERENCES:
- See also: Full FDA approved prescribing information can be found here — http://www.novantrone.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Trial Initiation Date: 17 October 2000 (date of first subject first visit). Trial Completion Date 15 July 2008 (date of last subject last visit). 46 centers enrolled at least one subject.
Groups:
- Novantrone Therapy: Novantrone, 12 mg/m2 intravenously once every 3 months, until a 140 mg/m2 cumulative dose was reached
Period: Overall Study
Arm/Group | Novantrone Therapy
Started | 509 (Patients with validated data who received at least 1 dose of Novantrone®)
Completed | 172 (Patients in the study for 5 years +/-3 months are considered to have completed the 5-year study)
Not Completed | 337
Not completed — Changing physicians | 38
Not completed — Death | 12
Not completed — Patient's decision | 92
Not completed — Other | 95
Not completed — Lost to Follow-up | 70
Not completed — Administrative withdrawal | 30

BASELINE CHARACTERISTICS:
Arm/Group | Novantrone Therapy
Number analyzed (Participants) | 509
Age, Customized [Number; unit: participants]
  <=18 years | 0
  18 - 70 years | 509
Age Continuous [Mean (Full Range); unit: years] | 46 [19 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 344
  Male | 165
Region of Enrollment [Number; unit: participants]
  United States | 509

OUTCOME MEASURES:

1. Primary Outcome: Congestive Heart Failure (Treatment Phase)
Description: Number of patients experiencing congestive heart failure during the treatment phase of the trial
Time Frame: up to 36 months
Measure: Number; unit: participants
Arm/Group | Novantrone Therapy
Number analyzed (Participants) | 509
participants | 6

2. Primary Outcome: Congestive Heart Failure (Annual Follow-Up Phase)
Description: Number of patients experiencing congestive heart failure during the annual follow-up phase of the trial
Time Frame: up to 5 years
Population: participants with annual follow up data
Measure: Number; unit: participants
Arm/Group | Novantrone Therapy
Number analyzed (Participants) | 250
participants | 4

3. Primary Outcome: Left Ventricular Ejection Fraction (Treatment Phase)
Description: Number of patients with left ventricular ejection fraction test results that decreased below 50% during the treatment phase of the trial
Time Frame: up to 36 months
Measure: Number; unit: participants
Arm/Group | Novantrone Therapy
Number analyzed (Participants) | 509
participants | 27

4. Primary Outcome: Left Ventricular Ejection Fraction (Annual Follow-Up Phase)
Description: Number of patients with left ventricular ejection fraction test results that decreased below 50% during the annual follow-up phase of the trial
Time Frame: up to 5 years
Population: participants with annual follow up data
Measure: Number; unit: participants
Arm/Group | Novantrone Therapy
Number analyzed (Participants) | 250
participants | 14

5. Primary Outcome: Serious Infections (Treatment Phase)
Description: Number of serious infections during the treatment phase of the trial
Time Frame: up to 36 months
Measure: Number; unit: number of infections
Arm/Group | Novantrone Therapy
Number analyzed (Participants) | 509
number of infections | 50

6. Primary Outcome: Serious Infections (Annual Follow-Up Phase)
Description: Number of serious infections during the annual follow-up phase of the trial
Time Frame: up to 5 years
Population: participants with annual follow up data
Measure: Number; unit: number of infections
Arm/Group | Novantrone Therapy
Number analyzed (Participants) | 250
number of infections | 0

7. Primary Outcome: IV Antibiotics (Individual Drugs Unspecified) Utilized Due to Serious Infection (Treatment Phase)
Description: Number of subjects in whom IV antibiotics were utilized due to serious infection during the treatment phase
Time Frame: up to 36 months
Measure: Number; unit: participants
Arm/Group | Novantrone Therapy
Number analyzed (Participants) | 509
participants | 40

8. Primary Outcome: IV Antibiotics (Individual Drugs Unspecified) Utilized Due To Serious Infection (Annual Follow-Up Phase)
Description: Number of subjects in whom IV antibiotics were utilized due to serious infection during the annual follow-up phase
Time Frame: up to 5 years
Population: participants with annual follow up data
Measure: Number; unit: participants
Arm/Group | Novantrone Therapy
Number analyzed (Participants) | 250
participants | 0

9. Primary Outcome: Severe Neutropenia (Treatment Phase)
Description: Number of infections associated with severe neutropenia at onset during the treatment phase
Time Frame: up to 36 months
Measure: Number; unit: number of infections
Arm/Group | Novantrone Therapy
Number analyzed (Participants) | 509
number of infections | 9

10. Primary Outcome: Severe Neutropenia (Annual Follow-Up Phase)
Description: Number of infections associated with severe neutropenia at onset during the annual follow-up phase
Time Frame: up to 5 years
Population: participants with annual follow up data
Measure: Number; unit: number of infections
Arm/Group | Novantrone Therapy
Number analyzed (Participants) | 250
number of infections | 0

11. Primary Outcome: Clinical Relapses (Treatment Phase)
Description: Number of clinical relapses reported during the treatment phase of the trial
Time Frame: up to 36 months
Measure: Number; unit: number of relapses
Arm/Group | Novantrone Therapy
Number analyzed (Participants) | 509
number of relapses | 185

12. Primary Outcome: Clinical Relapses (Annual Follow-Up Phase)
Description: Number of clinical relapses reported during the annual follow-up phase of the trial
Time Frame: up to 5 years
Population: participants with annual follow up data
Measure: Number; unit: number of relapses
Arm/Group | Novantrone Therapy
Number analyzed (Participants) | 250
number of relapses | 60

13. Primary Outcome: Symptomatic CHF, Left Ventricular Ejection Fraction - Prior to Each Dose • Serious Infections, IV Antibiotics, or Assoc w/ Severe Neutropenia-evaluated. Novantrone Admin - Per PI • SAE, Clinical Relapses
Description: Outcomes are presented separately above apart from adverse events which are presented in the adverse event section
Time Frame: up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 5 years. Combined serious adverse events are displayed for both the Treatment Phase and Annual Follow-Up Phase
Description: Only serious adverse events were collected in this study
Arm/Group | Novantrone Therapy
Serious Adverse Events (participants affected / at risk) | 102/509
Other Adverse Events (participants affected / at risk) | 0/509
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Novantrone Therapy (N=509)
Urinary Tract Infection (Infections and infestations) | 13 (17)
Pneumonia (Infections and infestations) | 5 (8)
Urosepsis (Infections and infestations) | 4 (4)
Cellulitis (Infections and infestations) | 3 (3)
Sepsis (Infections and infestations) | 3 (3)
Lobar Pneumonia (Infections and infestations) | 2 (2)
Shock Septic (Infections and infestations) | 2 (2)
Viral Infection (Infections and infestations) | 2 (2)
Bronchitis Viral (Infections and infestations) | 1 (1)
Cellulitis Gangrenous (Infections and infestations) | 1 (1)
Cystitis (Infections and infestations) | 1 (1)
Fungal Skin Infection (Infections and infestations) | 1 (1)
Herpes Zoster (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Localised Infection (Infections and infestations) | 1 (1)
Lung Infection (Infections and infestations) | 1 (1)
Meningitis (Infections and infestations) | 1 (1)
Postoperative Wound Infection (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1)
Urinary Tract Infection Enterococcal (Infections and infestations) | 1 (1)
Varicella (Infections and infestations) | 1 (1)
Wound Sepsis (Infections and infestations) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 5 (5)
Myocardial Infarction (Cardiac disorders) | 4 (4)
Cardiac Failure Congestive (Cardiac disorders) | 2 (2)
Tachycardia (Cardiac disorders) | 2 (2)
Cardio-respiratory Arrest (Cardiac disorders) | 1 (1)
Mitral Valve Incompetence (Cardiac disorders) | 1 (1)
Ventricular Hypokinesia (Cardiac disorders) | 1 (1)
Ejection Fraction Decreased (Investigations) | 14 (14)
Methicilin-resistant Staphylococcal Aureus Test Positive (Investigations) | 1 (1)
Road Traffic Accident (Injury, poisoning and procedural complications) | 4 (4)
Hip Fracture (Injury, poisoning and procedural complications) | 2 (2)
Fibula Fracture (Injury, poisoning and procedural complications) | 1 (1)
Humerus Fracture (Injury, poisoning and procedural complications) | 1 (1)
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 1 (1)
Rib Fracture (Injury, poisoning and procedural complications) | 1 (1)
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 (1)
Tendon Rupture (Injury, poisoning and procedural complications) | 1 (1)
Tibia Fracture (Injury, poisoning and procedural complications) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (3)
Fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal Disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Grand Mal Convulsion (Nervous system disorders) | 2 (2)
Muscle Spasticity (Nervous system disorders) | 2 (2)
Carotid Artery Occlusion (Nervous system disorders) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Transient Ischemic Attack (Nervous system disorders) | 1 (1)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Acute Myeloid Leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Acute Promyelocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Chronic Myeloid Leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Endometrial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pituitary Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 6 (6)
Hypertension (Vascular disorders) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 3 (3)
Abdominal Pain (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Depression (Psychiatric disorders) | 2 (2)
Major Depression (Psychiatric disorders) | 1 (1)
Mental Status Changes (Psychiatric disorders) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 1 (1)
Drug Delivery Device Implantation (Surgical and medical procedures) | 4 (4)
Medical Device Implantation (Surgical and medical procedures) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Chest Pain (General disorders) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 2 (2)
Hypothyroidism (Endocrine disorders) | 1 (1)
Anaphylactoid Reaction (Immune system disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Abortion Incomplete (Pregnancy, puerperium and perinatal conditions) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other